CLINICAL TRIAL: NCT02100514
Title: A 52 Week Phase 3 Double-blind, Randomized, Placebo-controlled, Parallel-group Study To Assess The Efficacy, Safety And Tolerability Of Pf-04950615 In Subjects With Primary Hyperlipidemia Or Mixed Dyslipidemia At Risk Of Cardiovascular Events
Brief Title: Randomized Clinical Trial of Bococizumab (PF-04950615; RN316) in Subjects With Primary Hyperlipidemia or Mixed Dyslipidemia At Risk Of Cardiovascular Events
Acronym: SPIRE-LL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1481045; SPIRE-LL (Other: Alias Study Number); 2014-000478-20 (EudraCT Number)
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Hyperlipidemia
Keywords: Primary hyperlipidemia or mixed dyslipidemia; high risk of cardiovascular events; multiple cardiovascular disease risk factors.
MeSH Terms: conditions — Hyperlipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bococizumab (PF-04950615; RN316) (Experimental): Bococizumab (PF-04950615; RN316)
  Interventions: Drug: Bococizumab (PF-04950615; RN316)
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bococizumab (PF-04950615; RN316) — 150 mg every 2 weeks, subcutaneous injection for 52 weeks.
  Arms: Bococizumab (PF-04950615; RN316)
Other: Placebo — Subcutaneous injection every 2 weeks for 52 weeks.
  Arms: placebo

SUMMARY:
This study is a multicenter, double-blind, randomized study to access the efficacy, safety and tolerability of Bococizumab (PF-04950615; RN316) in subjects with hyperlipidemia receiving background statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Treated with a statin
* Fasting LDL-C >=100 mg/dL and triglyceride <= 400 mg/dL
* High or very high risk of incurring a cardiovascular event

Exclusion Criteria:

* Pregnant or breastfeeding females
* Cardiovascular or cerebrovascular event or procedure within 90 days
* Congestive heart failure NYHA class IV
* Poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (222):
- United States (107):
  - Advanced Cardiovascular, LLC Research, Alexander City, Alabama
  - Advanced Cardiovascular, LLC, Research, Auburn, Alabama
  - Clinical Research Advantage, Inc./Family Practice Specialists, Ltd., Phoenix, Arizona
  - Clinical Research Advantage, Inc./Family Practice Specialists, LTD, Phoenix, Arizona
  - Radiant Research, Inc., Tucson, Arizona
  - Radiant Research, Inc, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - The Office of Larry Watkins, MD, Little Rock, Arkansas
  - American Institute of Research, Los Angeles, California
  - lntermed Group, Los Angeles, California
  - IMD Medical Group, Los Angeles, California
  - The Office of Lucita M. Cruz, M.D., Inc., Norwalk, California
  - Superior Research, LLC, Sacramento, California
  - Superior Research ,LLC, Sacramento, California
  - Radiant Research, Inc., Santa Rosa, California
  - Orange County Research Center, Tustin, California
  - Ventura Clinical Trials, Ventura, California
  - University of Colorado Hospital, Aurora, Colorado
  - Clinical Research Advantage, Inc. / Colorado Springs Family Practice, Colorado Springs, Colorado
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Boca Raton Clinical Research Associates, Boca Raton, Florida
  - BRCR Medical Center, Inc., Boca Raton, Florida
  - Meridien Research, Brooksville, Florida
  - Linfritz Research Institute Inc., Coral Gables, Florida
  - Florida Health Center, Fort Lauderdale, Florida
  - Health Care Family Rehab & Research Center, Hialeah, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Sunrise Research Institute, Inc, Miami, Florida
  - Prestige Clinical Research Center, Inc., Miami, Florida
  - Suncoast Research Group, LLD, Miami, Florida
  - Elite Clinical Research, Miami, Florida
  - Advanced Clinical Research of Miami, Miami, Florida
  - The Research Specialists of Florida, Inc., Miami, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - NewPhase Clinical Trials, Corp., Miami Beach, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Precision Research Organization, Miami Lakes, Florida
  - First Quality, Miramar, Florida
  - American Family Medical, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Andres Patron, D.O.P.A., Pembroke Pines, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Accord Clinical Research, Llc, Port Orange, Florida
  - East Coast Institute for Research, LLC/ Baker-Gilmour Cardiovascular Institute, Saint Augustine, Florida
  - East Coast Institute for RSCH, St. Augustine Cardiology Associates, Research, Saint Augustine, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Northwest Clinical Trials, Inc., Boise, Idaho
  - American Health Network of Indiana, LLC, Avon, Indiana
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Northwest Family Physicians, Wichita, Kansas
  - Imperial Health, LLP, Lake Charles, Louisiana
  - Crescent City Clinical Research Center, LLC, Metairie, Louisiana
  - Clinical Trials of America LA, Monroe, Louisiana
  - Bethesda Health Research, Bethesda, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - McLaren Flint, Flint, Michigan
  - CentraCare Heart & Vascular Center @ St. Cloud Hospital, Saint Cloud, Minnesota
  - CentraCare Heart & Vascular Center at St. Cloud Hospital, Saint Cloud, Minnesota
  - Riser Medical Research, Picayune, Mississippi
  - Washington University, The Center for Advanced Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Clinical Research Advantage, Inc. (Prairie Fields Family Medicine, PC), Fremont, Nebraska
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Physician's East Endocrinology, Greenville, North Carolina
  - Physician's East P.A., Greenville, North Carolina
  - Physician's East, PA, Greenville, North Carolina
  - Catawba Valley Medical Group, Inc., Hickory, North Carolina
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - PMG Research of Hickory, Hickory, North Carolina
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Primed Clinical Research, Dayton, Ohio
  - Office of Daniel G. Williams, MD, Perrysburg, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Consultants,LLC, Tulsa, Oklahoma
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - Medical Research South, LLC, Charleston, South Carolina
  - Ellipsis Research Group, LLC, Columbia, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Stern Cardiovascular Foundation, Inc, Germantown, Tennessee
  - Apex Cardiology, Jackson, Tennessee
  - Research Associates of Jackson, Jackson, Tennessee
  - PMG Research, Inc d/b/a PMG Research of Knoxville, Knoxville, Tennessee
  - Punzi Medical Center, Carrollton, Texas
  - Juno Research, LLC, Houston, Texas
  - Gulf Coast Medical Research,LLC, Houston, Texas
  - Office of Michelle Zaniewski MD., PA., Houston, Texas
  - Juno Research, LLC, Katy, Texas
  - Gulf Coast Medical Research, LLC, Missouri City, Texas
  - Clinical Research Advantage, Inc./ Plano Internal Medicine Associates, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Gulf Coast Medical Research, LLC, Sugar Land, Texas
  - Aspen Clinical Research, Orem, Utah
  - Millennium Clinical Trials, LLC, Arlington, Virginia
  - National Clinical Research-Norfolk, Inc., Norfolk, Virginia
  - Sound Health Care Center, Port Orchard, Washington
  - Sound Medical Research, Port Orchard, Washington
  - Walla Walla Clinic, Walla Walla, Washington
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
  - HFM Heart and Vascular Center/Holy Family Memorial, Inc, Manitowoc, Wisconsin
- Canada (33):
  - LMC Clinical Research Inc. (Calgary), Calgary, Alberta
  - Office of Dr. Ronald Collette MD, Burnaby, British Columbia
  - Medical Arts Health Research Group, Kamloops, British Columbia
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Glover Medical Clinic, Langley, British Columbia
  - Fraser Clinical Trials, New Westminster, British Columbia
  - The Medical Arts Health Research Group, Penticton, British Columbia
  - The Office of James K. Lai, MD Inc., Vancouver, British Columbia
  - Cook Street Medical Clinic, Victoria, British Columbia
  - LMC Clinical Research Inc. (Barrie), Barrie, Ontario
  - LMC Clinical Research Inc. (Brampton), Brampton, Ontario
  - Aggarwal And Associates Ltd, Brampton, Ontario
  - Corunna Medical Research Centre, Corunna, Ontario
  - LMC Clinical Research Inc. (Etobicoke), Etobicoke, Ontario
  - LMC Clinical Research Inc. (Markham), Markham, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - LMC Clinical Research Inc. (Oakville), Oakville, Ontario
  - The Office of Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - LMC Clinical Research Inc. (Thornhill), Thornhill, Ontario
  - Rouge Valley Health System - Centenary, Toronto, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - Manna Research Inc., Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - ViaCar Recherche Clinique Inc., Greenfield Park, Quebec
  - Centre de Depistage et de Recherche Cardiovasculaire Rive-Sud, Longueuil, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Clinique des maladies lipidiques de Quebec, Québec, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
  - Centre De Sante Et De Services Sociaux De Beauce (CSSSB), Saint-Georges, Beauce, Quebec
  - C.I.C. Maurice Inc., Trois-Rivières, Quebec
  - C.I.C. Mauricie Inc., Trois-Rivières, Quebec
- Czechia (20):
  - Kardiologicka ambulance, Trutnov, Královéhradecký kraj
  - Fakultni Nemocnice Kralovske Vinohrady, II. interni klinika, Prague, Vinohrady
  - Fakultni nemocnice u sv. Anny Brno. Oddeleni klinicke biochemie, Brno
  - Fakultni nemocnice u sv. Anny. Nemoenicni lekarna (pharmacy), Brno
  - Cardiocentrum Kladno s.r.o., Kardiologicka ambulance, Kladno
  - Lekarna - P-P Klinika Kladno, Kladno
  - Lunacor s.r.o., Kroměříž
  - Fakultni Nemocnice Olomouc, III. interni klinika ¿ nefrologicka, revmatologicka a endokrinologicka, Olomouc
  - Lekarna Fakultni nemocnice Olomouc (pharmacy), Olomouc
  - Lekarna Domovina, Olomouc
  - PreventaMed, s.r.o., Olomouc
  - IKEM, Oddeleni preventivni kardiologie, Prague
  - IKEM, Ustavni lekarna, Prague
  - BENU lekarna, Příbram
  - Kardiologicka ambulance, III. Poliklinika, Příbram
  - Lekarna 203-02, Slaný
  - Nemocnice Slany, Interni oddeleni, Slaný
  - AeskuLab k.s., Lipidova poradna, Teplice
  - Lekarna Centrum (pharmacy), Teplice
  - Dr.Max lekarna, Trutnov
- Finland (2):
  - Etela-Karjalan Keskussairaala, Lappeenranta
  - Turku University Hospital, Turku
- Netherlands (13):
  - Medisch Spectrum Twente, Enschede, ER
  - St Lucas Andreas Hospital, Amsterdam, North Holland
  - Gelre Hospitals, Apeldoorn
  - Andromed Eindhoven, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Beatrix Hospital, Gorinchem
  - Martini Ziekenhuis, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Andro Medical Research B.V., Rotterdam
  - Ikazia Hospital, Rotterdam
  - D&A Research and Genetics, Sneek
  - St. Elisabeth Hospital, Tilburg
  - University Medical Center Utrecht, Utrecht
- Norway (3):
  - Ossum Gronert Legetjeneste AS, Hønefoss
  - Oslo Universitetssykehus HF, Oslo
  - Oslo Universitetssykehus HF, Ulleval, Oslo
- Poland (15):
  - KO-MED Centra Kliniczne Lublin, Lublin, Lublin Voivodeship
  - KO-MED Centra Kliniczne Zamosc, Zamość, Lublin Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - MCBK Sc lwona Czajkowska Monika Barney, Grodzisk Mazowiecki
  - Synexus Polska Sp. z o. o. Oddizial w Katowicach., Katowice
  - Clinport Tura Lipinska Dabrowski S.C., Katowice
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Jan Zbigniew Peruga NZOZ SALUS, Lodz
  - Zespol Opieki Zdrowotnej W Olawie, Oddzial Chorob Wewnetrznych, Oława
  - Synexus Polska Sp. z o.o Oddzial w Poznaniu, Poznan
  - KO-MED Centra Kliniczne Sp. z o.o., Puławy
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
  - .WroMedica Irena Bielicka, Janusz Szczepanik Spolka Cywlina, Wroclaw
  - KO-MED. Centra Kliniczne Staszow, Staszów, Świętokrzyskie Voivodeship
- Puerto Rico (3):
  - Ponce School Of Medicine, Ponce, PR
  - Cardiometabolic Research Center, Inc, Ponce, PR
  - Caparra Internal Medicine, Río Grande
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore
- South Korea (4):
  - Sacred Heart Hospital-Hallym University, Anyang-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Sweden (8):
  - Clinical Trial Center (CTC)/Centrum foer klinisk proevning, Gothenburg
  - Vardcentralen Lessebo, Lessebo
  - Clinical Trials Consultants AB, Linköping
  - ProbarE i Lund AB, Lund
  - Capio Citykliniken Hjartmottagning, Lund
  - Dalecarlia Clinical Research Center, Rättvik
  - Citydiabetes, Stockholm
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- United Kingdom (12):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berkshire
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - Synexus Scotland Clinical Research Centre, Glasgow, Lanarkshire Scotland
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - Synexus North East Clinical Research Centre - Hexham General Hospital, Hexham, Northumberland
  - Worcestershire Acute Hospitals NHS Trust - Worcestershire Royal Hospital, Worcester, Worcestershire
  - University Hospital Ayr - Nhs Ayrshire And Arran, Ayr
  - Synexus Midlands Clinical Research Centre, Birmingham
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Synexus Merseyside Clinical Research Centre, Liverpool
  - Synexus Manchester Clinical Research Centre, Manchester
  - Abertawe Bro Morgannwg University Local Health Board Joint Clinical Research Facility,, Swansea

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] McCush F, Wang E, Yunis C, Schwartz P, Baltrukonis D. Anti-drug Antibody Magnitude and Clinical Relevance Using Signal to Noise (S/N): Bococizumab Case Study. AAPS J. 2023 Sep 2;25(5):85. doi: 10.1208/s12248-023-00846-x. PMID 37658997
- [Derived] Chasman DI, Hyde CL, Giulianini F, Danning RD, Wang EQ, Hickling T, Ridker PM, Loomis AK. Genome-wide pharmacogenetics of anti-drug antibody response to bococizumab highlights key residues in HLA DRB1 and DQB1. Sci Rep. 2022 Mar 11;12(1):4266. doi: 10.1038/s41598-022-07997-5. PMID 35277540
- [Derived] Ridker PM, Rose LM, Kastelein JJP, Santos RD, Wei C, Revkin J, Yunis C, Tardif JC, Shear CL; Studies of PCSK9 Inhibition and the Reduction of vascular Events (SPIRE) Investigators. Cardiovascular event reduction with PCSK9 inhibition among 1578 patients with familial hypercholesterolemia: Results from the SPIRE randomized trials of bococizumab. J Clin Lipidol. 2018 Jul-Aug;12(4):958-965. doi: 10.1016/j.jacl.2018.03.088. Epub 2018 Apr 3. PMID 29685591
- [Derived] Ridker PM, Tardif JC, Amarenco P, Duggan W, Glynn RJ, Jukema JW, Kastelein JJP, Kim AM, Koenig W, Nissen S, Revkin J, Rose LM, Santos RD, Schwartz PF, Shear CL, Yunis C; SPIRE Investigators. Lipid-Reduction Variability and Antidrug-Antibody Formation with Bococizumab. N Engl J Med. 2017 Apr 20;376(16):1517-1526. doi: 10.1056/NEJMoa1614062. Epub 2017 Mar 17. PMID 28304227
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481045&StudyName=Randomized%20Clinical%20Trial%20of%20RN316%20%28PF-04950615%29%20inSubjects%20With%20Primary%20Hyperlipidemia%20or%20Mixed%20Dyslipidemia%20At%20Risk%20Of%20Cardiovascular%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at multiple sites from 28 October 2014 to 15 July 2016 for the treatment period and up to 10 July 2017 for the extension period.
Groups:
- Treatment Period: Placebo: Participants received placebo matched to Bococizumab (PF-04950615) subcutaneous injection once every 2 weeks up to Week 52. Participants were followed up to Week 58.
- Treatment Period: Bococizumab 150 mg: Participants received Bococizumab (PF-04950615) 150 milligram (mg) subcutaneous injection once every 2 weeks up to Week 52. Participants were followed up to Week 58.
- Extension Period: Placebo: Participants randomized to Placebo arm in treatment period and consented for extension period after Week 58 follow-up visit, were followed for SAEs and concomitant medications up to Week 110.
- Extension Period: Bococizumab ADA Positive: Participants randomized to Bococizumab in treatment period were classified as either ADA positive or ADA negative based on their ADA assessment at Week 58 follow-up visit. In extension period, participants who were ADA positive and consented for extension period were assessed for ADA and LDL-C direct measurement until ADA titers were no longer detectable or had returned to baseline titer (less than or equal to 1.58 (log2) units above a positive baseline titer) or until Week 110 along with SAEs and concomitant medication, from Week 58 follow up visit to Week 110.
- Extension Period: Bococizumab ADA Negative: Participants randomized to Bococizumab in treatment period were classified as either ADA positive or ADA negative based on their Week 58 follow-up ADA assessment. Participants who were ADA negative and consented for extension period were followed for SAEs and concomitant medication, from Week 58 follow up visit to Week 110.
Period: Treatment Period
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg | Extension Period: Placebo | Extension Period: Bococizumab ADA Positive | Extension Period: Bococizumab ADA Negative
Started | 247 | 499 | 0 | 0 | 0
Completed | 218 | 425 | 0 | 0 | 0
Not Completed | 29 | 74 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 5 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 17 | 0 | 0 | 0
Not completed — Did Not Meet Entrance Criteria | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 37 | 0 | 0 | 0
Not completed — Other | 9 | 11 | 0 | 0 | 0
Period: Extension Period
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg | Extension Period: Placebo | Extension Period: Bococizumab ADA Positive | Extension Period: Bococizumab ADA Negative
Started | 0 | 0 | 44 | 33 | 56
Completed | 0 | 0 | 42 | 33 | 56
Not Completed | 0 | 0 | 2 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized.
Groups:
- Treatment Period: Bococizumab 150 mg: Participants received Bococizumab (PF-04950615) 150 mg subcutaneous injection once every 2 weeks up to Week 52. Participants were followed up to Week 58.
- Total: Total of all reporting groups
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg | Total
Number analyzed (Participants) | 247 | 499 | 746
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.0) | 61.5 (9.9) | 61.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 223 | 330
  Male | 140 | 276 | 416

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: FAS included all participants who were randomized. Here, "Number of participants analyzed (N)" signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 235 | 468
percent change | -0.8 (17.61) | -50.8 (29.81)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Least square (LS) mean difference and associated 95% confidence interval (CI), and p-value were derived from an mixed effect model repeat measurement (MMRM) model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference compared to placebo = -49.9, 95% CI 2-sided [-54.0 to -45.8], Standard Error of Mean 2.09

2. Secondary Outcome: Percent Change From Baseline in Fasting Total Cholesterol (TC) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, "n" signifies number of participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 236 | 469
  Week 12 | -2.2 (13.41) | -35.4 (20.93)
  Week 24: number analyzed (Participants) | 237 | 463
  Week 24 | -3.1 (15.79) | -32.9 (23.06)
  Week 52: number analyzed (Participants) | 221 | 425
  Week 52 | -5.0 (17.22) | -29.0 (22.08)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 12: LS mean difference and associated 95% CI and p-value were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference compared to placebo = -33.2, 95% CI 2-sided [-36.1 to -30.2], Standard Error of Mean 1.48
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 24: LS mean difference and associated 95% CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -29.6, 95% CI 2-sided [-32.8 to -26.3], Standard Error of Mean 1.66
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 52: LS mean difference and associated 95% CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -23.8, 95% CI 2-sided [-27.0 to -20.5], Standard Error of Mean 1.65

3. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein B (ApoB) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 234 | 467
  Week 12 | -0.6 (16.70) | -46.5 (28.87)
  Week 24: number analyzed (Participants) | 236 | 461
  Week 24 | -2.1 (18.66) | -43.5 (32.26)
  Week 52: number analyzed (Participants) | 221 | 425
  Week 52 | -4.4 (20.77) | -37.3 (29.59)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 12: LS mean difference and associated 95% CI, and p-value were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference compared to placebo = -45.7, 95% CI 2-sided [-49.7 to -41.7], Standard Error of Mean 2.04
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 24: LS mean difference and associated 95% CI, were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -40.9, 95% CI 2-sided [-45.3 to -36.5], Standard Error of Mean 2.26
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 52: LS mean difference and associated 95% CI, were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -32.5, 95% CI 2-sided [-36.7 to -28.2], Standard Error of Mean 2.17

4. Secondary Outcome: Percent Change From Baseline in Fasting Non High Density Lipoprotein Cholesterol (Non HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 236 | 469
  Week 12 | -2.6 (17.57) | -47.6 (28.36)
  Week 24: number analyzed (Participants) | 237 | 463
  Week 24 | -3.8 (20.63) | -44.7 (30.83)
  Week 52: number analyzed (Participants) | 221 | 425
  Week 52 | -6.4 (22.70) | -39.5 (29.36)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference compared to placebo = -45.0, 95% CI 2-sided [-48.9 to -41.1], Standard Error of Mean 1.99
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 24: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -40.5, 95% CI 2-sided [-44.8 to -36.1], Standard Error of Mean 2.21
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 52: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -32.7, 95% CI 2-sided [-37.0 to -28.4], Standard Error of Mean 2.20

5. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) by Triglycerides Cut-off of Less Than (<) 200 Milligram Per Deciliter (mg/dL) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: A subset of FAS included all participants who were randomized and had TG <200 mg/dL at pre-randomization. Here, "n" signifies number of participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 164 | 331
percent change
  Week 12: number analyzed (Participants) | 158 | 313
  Week 12 | 0.5 (16.61) | -51.1 (30.43)
  Week 24: number analyzed (Participants) | 159 | 311
  Week 24 | -1.6 (21.68) | -48.4 (33.67)
  Week 52: number analyzed (Participants) | 148 | 292
  Week 52 | -4.2 (24.11) | -42.2 (33.75)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 12: LS mean difference and associated 95% CI and p-value were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference compared to placebo = -51.6, 95% CI 2-sided [-56.7 to -46.6], Standard Error of Mean 2.59
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 24: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -46.4, 95% CI 2-sided [-52.2 to -40.6], Standard Error of Mean 2.94
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 52: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -37.4, 95% CI 2-sided [-43.3 to -31.4], Standard Error of Mean 3.03

6. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) by Triglycerides Cut-off of Greater Than or Equal to (>=) 200 Milligram Per Deciliter (mg/dL) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: A subset of FAS included all participants who were randomized and had TG >=200 mg/dL at pre-randomization. Here, "n" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 83 | 168
percent change
  Week 24: number analyzed (Participants) | 77 | 150
  Week 24 | -5.7 (21.67) | -45.8 (33.13)
  Week 52: number analyzed (Participants) | 74 | 133
  Week 52 | -5.7 (23.78) | -40.9 (30.25)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference compared to placebo = -46.6, 95% CI [-53.7 to -39.5], Standard Error of Mean 3.59
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 24: LS mean difference and associated 95% CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -39.7, 95% CI [-47.9 to -31.6], Standard Error of Mean 4.12
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 52: LS mean difference and associated 95% CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -33.4, 95% CI [-41.3 to -25.5], Standard Error of Mean 4.02

7. Secondary Outcome: Percent Change From Baseline in Fasting Lipoprotein (A) (Lp[A]) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 235 | 469
  Week 12 | 4.9 (54.24) | -25.7 (29.45)
  Week 24: number analyzed (Participants) | 235 | 463
  Week 24 | 5.9 (50.52) | -21.3 (34.42)
  Week 52: number analyzed (Participants) | 221 | 425
  Week 52 | 27.9 (374.64) | -21.5 (32.61)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference compared to placebo = -30.8, 95% CI [-36.9 to -24.6], Standard Error of Mean 3.14
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; LS mean difference compared to placebo = -27.5, 95% CI [-33.9 to -21.2], Standard Error of Mean 3.23
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; LS mean difference compared to placebo = -49.4, 95% CI 2-sided [-85.2 to -13.5], Standard Error of Mean 18.27

8. Secondary Outcome: Percent Change From Baseline in Fasting High Density Lipoprotein Cholesterol (HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, "n" signifies number of participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 236 | 469
  Week 12 | 0.6 (13.93) | 6.3 (13.86)
  Week 24: number analyzed (Participants) | 237 | 463
  Week 24 | 0.6 (14.88) | 6.3 (14.49)
  Week 52: number analyzed (Participants) | 221 | 425
  Week 52 | 0.7 (14.24) | 7.0 (15.60)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference compared to placebo = 5.5, 95% CI 2-sided [3.4 to 7.6], Standard Error of Mean 1.06
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; LS mean difference compared to placebo = 5.4, 95% CI [3.2 to 7.6], Standard Error of Mean 1.14
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; LS mean difference compared to placebo = 6.0, 95% CI [3.6 to 8.3], Standard Error of Mean 1.20

9. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 24, 52: Treatment Period
Time Frame: Baseline, Week 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 24: number analyzed (Participants) | 236 | 461
  Week 24 | -2.9 (21.72) | -47.5 (33.48)
  Week 52: number analyzed (Participants) | 222 | 425
  Week 52 | -4.7 (23.96) | -41.8 (32.67)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; LS mean difference compared to placebo = -44.2, 95% CI [-48.8 to -39.5], Standard Error of Mean 2.39
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; LS mean difference compared to placebo = -36.2, 95% CI 2-sided [-40.9 to -31.4], Standard Error of Mean 2.42

10. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 236 | 469
  Week 12 | -6.2 (32.92) | -16.2 (32.86)
  Week 24: number analyzed (Participants) | 237 | 463
  Week 24 | -8.9 (35.60) | -18.2 (65.13)
  Week 52: number analyzed (Participants) | 221 | 425
  Week 52 | -8.0 (41.46) | -15.8 (35.57)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 12: LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -10.1, 95% CI [-15.1 to -5.1], Standard Error of Mean 2.55
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; LS mean difference compared to placebo = -9.0, 95% CI [-17.9 to -0.2], Standard Error of Mean 4.50
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; LS mean difference compared to placebo = -8.2, 95% CI [-14.1 to -2.2], Standard Error of Mean 3.04

11. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A-I (ApoA-I) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 236 | 468
  Week 12 | -0.9 (11.09) | 3.4 (11.43)
  Week 24: number analyzed (Participants) | 236 | 461
  Week 24 | -1.6 (10.81) | 2.5 (11.61)
  Week 52: number analyzed (Participants) | 221 | 425
  Week 52 | -1.0 (13.12) | 3.4 (11.77)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = 4.1, 95% CI [2.5 to 5.8], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; LS mean difference compared to placebo = 3.8, 95% CI [2.2 to 5.5], Standard Error of Mean 0.86
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; LS mean difference compared to placebo = 4.3, 95% CI [2.4 to 6.2], Standard Error of Mean 0.97

12. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A-II (ApoA-II) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 235 | 468
  Week 12 | 2.0 (11.94) | 3.0 (11.94)
  Week 24: number analyzed (Participants) | 233 | 462
  Week 24 | 2.6 (12.12) | 3.7 (14.12)
  Week 52: number analyzed (Participants) | 220 | 423
  Week 52 | 0.7 (12.46) | 1.9 (12.22)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = 1.1, 95% CI [-0.7 to 2.8], Standard Error of Mean 0.90
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; LS mean difference compared to placebo = 0.9, 95% CI [-1.1 to 3.0], Standard Error of Mean 1.04
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; LS mean difference compared to placebo = 0.8, 95% CI [-1.0 to 2.7], Standard Error of Mean 0.95

13. Secondary Outcome: Percent Change From Baseline in Fasting Very Low Density Lipoprotein Cholesterol (VLDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percent change
  Week 12: number analyzed (Participants) | 236 | 469
  Week 12 | -6.2 (32.92) | -16.2 (32.86)
  Week 24: number analyzed (Participants) | 237 | 463
  Week 24 | -8.9 (35.60) | -18.2 (65.13)
  Week 52: number analyzed (Participants) | 221 | 425
  Week 52 | -8.0 (41.46) | -15.8 (35.57)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = -10.1, 95% CI [-15.1 to -5.1], Standard Error of Mean 2.55
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; LS mean difference compared to placebo = -9.0, 95% CI [-17.9 to -0.2], Standard Error of Mean 4.50
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; LS mean difference compared to placebo = -8.2, 95% CI [-14.1 to -2.2], Standard Error of Mean 3.04

14. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) by Triglycerides Cut-off of Less Than (<) 200 Milligram Per Deciliter (mg/dL) at Week 12
Time Frame: Baseline, Week 12
Population: A subset of FAS included all participants who were randomized and had TG <200 mg/dL at pre-randomization. Here, "n" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 164 | 331
mg/dL
  Baseline | 130.1 (25.22) | 130.2 (28.72)
  Change at Week 12: number analyzed (Participants) | 158 | 313
  Change at Week 12 | -0.5 (22.37) | -67.3 (40.14)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction and geographical region. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -66.8, 95% CI [-73.0 to -60.5], Standard Error of Mean 3.18

15. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) by Triglycerides Cut-off of Greater Than or Equal to (>=) 200 Milligram Per Deciliter (mg/dL) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 83 | 168
mg/dL
  Baseline | 143.7 (35.49) | 147.2 (39.48)
  Change at Week 12: number analyzed (Participants) | 77 | 155
  Change at Week 12 | -6.6 (29.61) | -74.1 (48.04)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = -66.1, 95% CI [-76.7 to -55.4], Standard Error of Mean 5.40

16. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
mg/dL
  Baseline | 134.7 (29.71) | 135.9 (33.67)
  Change at Week 12: number analyzed (Participants) | 235 | 468
  Change at Week 12 | -2.5 (25.07) | -69.6 (42.98)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; LS mean difference and associated 95% CI were derived from MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -66.5, 95% CI [-72.0 to -61.1], Standard Error of Mean 2.77

17. Secondary Outcome: Absolute Change From Baseline in Fasting Total Cholesterol (TC) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
mg/dL
  Baseline | 209.4 (33.84) | 210.3 (37.97)
  Change at Week 12: number analyzed (Participants) | 236 | 469
  Change at Week 12 | -5.9 (29.61) | -75.4 (46.91)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = -69.1, 95% CI [-75.2 to -63.1], Standard Error of Mean 3.08

18. Secondary Outcome: Absolute Change From Baseline in Fasting Non High Density Lipoprotein Cholesterol (Non HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
mg/dL
  Baseline | 160.2 (33.49) | 162.1 (37.78)
  Change at Week 12: number analyzed (Participants) | 236 | 469
  Change at Week 12 | -5.8 (29.59) | -77.9 (48.28)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = -71.3, 95% CI [-77.5 to -65.1], Standard Error of Mean 3.14

19. Secondary Outcome: Absolute Change From Baseline in Fasting Apolipoprotein B (ApoB) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
mg/dL
  Baseline | 106.1 (20.43) | 107.1 (23.33)
  Change at Week 12: number analyzed (Participants) | 234 | 467
  Change at Week 12 | -1.6 (18.09) | -49.8 (31.81)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = -47.7, 95% CI [-51.9 to -43.6], Standard Error of Mean 2.12

20. Secondary Outcome: Absolute Change From Baseline in Fasting Lipoprotein (A) (Lp[A]) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
mg/dL
  Baseline | 48.5 (54.04) | 47.3 (53.55)
  Change at Week 12: number analyzed (Participants) | 235 | 469
  Change at Week 12 | 0.1 (10.91) | -10.3 (17.01)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = -10.4, 95% CI [-12.5 to -8.3], Standard Error of Mean 1.06

21. Secondary Outcome: Absolute Change From Baseline in Fasting High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
mg/dL
  Baseline | 49.2 (13.20) | 48.3 (11.60)
  Change at Week 12: number analyzed (Participants) | 236 | 469
  Change at Week 12 | -0.1 (6.75) | 2.5 (6.64)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = 2.6, 95% CI [1.6 to 3.6], Standard Error of Mean 0.52

22. Secondary Outcome: Absolute Change From Baseline in Ratio of Fasting Total Cholesterol (TC) to High Density Lipoprotein Cholesterol (HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
ratio
  Baseline | 4.6 (1.90) | 4.6 (1.31)
  Change at Week 12: number analyzed (Participants) | 236 | 469
  Change at Week 12 | -0.2 (1.27) | -1.8 (1.29)
  Change at Week 24: number analyzed (Participants) | 237 | 463
  Change at Week 24 | -0.2 (1.42) | -1.6 (1.38)
  Change at Week 52: number analyzed (Participants) | 221 | 425
  Change at Week 52 | -0.2 (1.62) | -1.5 (1.32)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; LS mean difference compared to placebo = -1.6, 95% CI [-1.8 to -1.5], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; LS mean difference compared to placebo = -1.4, 95% CI [-1.6 to -1.3], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; LS mean difference compared to placebo = -1.4, 95% CI [-1.6 to -1.2], Standard Error of Mean 0.12

23. Secondary Outcome: Absolute Change From Baseline in Ratio of Fasting Apolipoprotein B (ApoB) to Apolipoprotein A-I (ApoA-I) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, "n" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
ratio
  Baseline | 0.7 (0.25) | 0.8 (0.22)
  Change at Week 12: number analyzed (Participants) | 234 | 467
  Change at Week 12 | 0.0 (0.14) | -0.4 (0.25)
  Change at Week 24: number analyzed (Participants) | 236 | 461
  Change at Week 24 | -0.0 (0.16) | -0.3 (0.27)
  Change at Week 52: number analyzed (Participants) | 221 | 425
  Change at Week 52 | 0.0 (0.66) | -0.3 (0.25)
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 12: LS mean difference and associated 95% confidence interval CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -0.4, 95% CI [-0.4 to -0.3], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 24: LS mean difference and associated 95% confidence interval CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -0.3, 95% CI [-0.3 to -0.3], Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 52: LS mean difference and associated 95% confidence interval CI were derived from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region and triglyceride subgroup. An unstructured variance covariance matrix was used; Test type: Superiority or Other; LS mean difference compared to placebo = -0.3, 95% CI [-0.4 to -0.2], Standard Error of Mean 0.04

24. Secondary Outcome: Percentage of Participants Achieving Fasting Low Density Lipoprotein Cholesterol (LDL-C) Less Than or Equal to (<=) 100 Milligram Per Deciliter (mg/dL) at Week 12, 24 and 52
Time Frame: Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, 'n' signifies those participants who were evaluable at specified time points for each arm respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percentage of participants
  Week 12: number analyzed (Participants) | 235 | 468
  Week 12 | 10.2 | 81.6
  Week 24: number analyzed (Participants) | 236 | 461
  Week 24 | 19.9 | 75.1
  Week 52: number analyzed (Participants) | 222 | 425
  Week 52 | 25.2 | 72.7
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 12: Odds ratio, associated 95% CI were derived from a logistic regression model with fixed effects for treatment group, baseline value, geographical region and triglyceride subgroup; Test type: Superiority or Other; Odds Ratio (OR) = 53.9, 95% CI [32.08 to 90.59]
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 24: Odds ratio, associated 95% CI were derived from a logistic regression model with fixed effects for treatment group, baseline value, geographical region and triglyceride subgroup; Test type: Superiority or Other; Odds Ratio (OR) = 17.0, 95% CI [11.15 to 26.07]
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; Week 52: Odds ratio, associated 95% CI were derived from a logistic regression model with fixed effects for treatment group, baseline value, geographical region and triglyceride subgroup; Test type: Superiority or Other; Odds Ratio (OR) = 9.1, 95% CI [6.18 to 13.48]

25. Secondary Outcome: Percentage of Participants Achieving Fasting Low Density Lipoprotein Cholesterol (LDL-C) Less Than or Equal to (<=) 70 Milligram Per Deciliter (mg/dL) at Week 12, 24 and 52
Time Frame: Week 12, 24, 52
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
percentage of participants
  Week 12: number analyzed (Participants) | 235 | 468
  Week 12 | 1.3 | 62.2
  Week 24: number analyzed (Participants) | 236 | 461
  Week 24 | 1.7 | 60.1
  Week 52: number analyzed (Participants) | 222 | 425
  Week 52 | 3.2 | 53.4
Statistical Analysis 1: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 156.4, 95% CI [48.84 to 501.11]
Statistical Analysis 2: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 24, analysis 2]; Test type: Superiority or Other; Odds Ratio (OR) = 110.8, 95% CI [39.77 to 308.46]
Statistical Analysis 3: Comparison: Treatment Period: Placebo vs Treatment Period: Bococizumab 150 mg; [analysis description as in outcome 24, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 43.3, 95% CI [19.52 to 96.13]

26. Secondary Outcome: Plasma Concentration Versus Time Summary of PF-04950615
Time Frame: Week 12, 24, 52
Population: Analysis set included participants who received at least 1 dose of PF-04950615. This outcome measure was planned not to be analysed for placebo reporting arm. Here, "n" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 499
microgram per milliliter
  Week 12: number analyzed (Participants) | 456
  Week 12 | 5.37 (5.327)
  Week 24: number analyzed (Participants) | 448
  Week 24 | 5.28 (5.888)
  Week 52: number analyzed (Participants) | 418
  Week 52 | 4.01 (4.652)

27. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) Related to Type 1 and 3 Hypersensitivity Reactions and Injection Site Reactions
Description: Type 1 hypersensitivity or allergic reactions were possible in response to any injected protein and included shortness of breath, urticaria, anaphylaxis and angioedema. Type 3 hypersensitivity reactions were similar to Type 1 hypersensitivity reactions but were likely to be delayed from the time of injection and included symptoms such as rash, urticaria, polyarthritis, myalgia's, polysynovitis, fever and if severe then included glomerulonephritis. Injection site reactions included injection site bruising, discolouration, erythema, haematoma, haemorrhage, nodule, induration, inflammation, mass, pain, paraesthesia, pruritus, swelling, vesicles, warmth, scab and rash. Participants with type 1 or type 3 hypersensitivity reactions and participants with injection site reactions were reported in this outcome measure.
Time Frame: Baseline up to end of study (up to 110 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 247 | 499
Percentage of participants
  With type 1 or 3 hypersensitivity reactions | 0.0 | 0.2
  With injection site reactions | 0.8 | 13.4

28. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb): Treatment Period
Description: Percentage of participants with at least 1 positive ADA titer or 1 positive nAb titer were reported. ADA titer >=6.23 (log 2) unit was considered to be ADA positive and nAb titer >=1.58 (log 2) unit was considered to be nAb positive.
Time Frame: Baseline up to Week 58
Population: Analysis set included all participants who received at least 1 dose of PF-04950615 150 mg. This outcome measure was planned not to be analysed for placebo reporting arm. Here "N" signifies number of subjects who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Period: Bococizumab 150 mg
Number analyzed (Participants) | 491
Percentage of participants
  Baseline up to Week 58: ADA positive | 54.8
  Baseline up to Week 58: nAb positive | 37.9

29. Secondary Outcome: Number of Participants Who Changed Concomitant Medication During Extension Period
Description: In this outcome measure, total number of participants who changed their lipid-lowering medications or added a monoclonal antibody medication during the extension period were reported.
Time Frame: Week 58 follow-up to Week 110
Population: All participants who consented for extension period.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Period: Placebo | Extension Period: Bococizumab ADA Positive | Extension Period: Bococizumab ADA Negative
Number analyzed (Participants) | 44 | 33 | 56
Participants | 2 | 4 | 3

30. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 58 (Follow up), 71, 84, 97 and 110: Extension Period
Time Frame: Baseline, Week 58 (follow up), 71, 84, 97, 110
Population: All participants who consented for extension period. This outcome measure was planned not to be analyzed for reporting arms: Placebo (Extension Period) and Bococizumab ADA negative (Extension Period).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Extension Period: Bococizumab ADA Positive
Number analyzed (Participants) | 33
percent change
  Week 58 (follow up) | 6.7 (27.70)
  Week 71 | 8.7 (34.83)
  Week 84 | 7.0 (30.34)
  Week 97 | 2.6 (31.43)
  Week 110 | 15.5 (36.17)

31. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb): Extension Period
Description: Percentage of participants with at least 1 positive ADA titer or 1 positive nAb titer were reported. ADA titer >=6.23 log2 unit was considered to be ADA positive and nAb titer >=1.58 log2 unit was considered to be nAb positive.
Time Frame: Week 58 (follow-up), Week 71, Week 84, Week 97, Week 110
Population: All participants who consented for extension period. This outcome measure was planned not to be analyzed for reporting arms Placebo (Extension period) and Bococizumab ADA negative (Extension period). Here, "n" signifies number of participants who were evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Extension Period: Bococizumab ADA Positive
Number analyzed (Participants) | 33
percentage of participants
  Week 58 (follow up): ADA positive | 100.0
  Week 58 (follow up): nAB positive | 60.6
  Week 71: ADA positive: number analyzed (Participants) | 31
  Week 71: ADA positive | 87.1
  Week 71: nAB positive: number analyzed (Participants) | 31
  Week 71: nAB positive | 35.5
  Week 84: ADA positive: number analyzed (Participants) | 28
  Week 84: ADA positive | 82.1
  Week 84: nAB positive: number analyzed (Participants) | 28
  Week 84: nAB positive | 25.0
  Week 97: ADA positive: number analyzed (Participants) | 22
  Week 97: ADA positive | 86.4
  Week 97: nAB positive: number analyzed (Participants) | 22
  Week 97: nAB positive | 18.2
  Week 110: ADA positive: number analyzed (Participants) | 17
  Week 110: ADA positive | 100.0
  Week 110: nAB positive: number analyzed (Participants) | 17
  Week 110: nAB positive | 11.8

ADVERSE EVENTS:
Time Frame: For SAEs: Baseline up to Week 110 and for other AEs: Baseline up to Week 58
Description: Event may be serious in 1 and nonserious in other participant or 1 participant may have experienced both serious and nonserious AE. Participants evaluable:treatment period: participants who received at least 1 dose of study drug;extension period: participants who consented for extension period. Nonserious AEs were not collected for extension period.
Arm/Group | Treatment Period: Placebo | Treatment Period: Bococizumab 150 mg | Extension Period: Placebo | Extension Period: Bococizumab ADA Positive | Extension Period: Bococizumab ADA Negative
All-Cause Mortality (participants affected / at risk) | 2/247 | 2/499 | 0/44 | 0/33 | 0/56
Serious Adverse Events (participants affected / at risk) | 32/247 | 44/499 | 2/44 | 0/33 | 1/56
Other Adverse Events (participants affected / at risk) | 29/247 | 97/499 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: Placebo (N=247) | Treatment Period: Bococizumab 150 mg (N=499) | Extension Period: Placebo (N=44) | Extension Period: Bococizumab ADA Positive (N=33) | Extension Period: Bococizumab ADA Negative (N=56)
POSSIBLE SEIZURE DISORDER SECONDARY TO AMPHETAMINE ABUSE (General disorders) | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 3 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 4 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 5 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Vascular stent occlusion (General disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Miller Fisher syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral artery dissection (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: Placebo (N=247) | Treatment Period: Bococizumab 150 mg (N=499) | Extension Period: Placebo (N=0) | Extension Period: Bococizumab ADA Positive (N=0) | Extension Period: Bococizumab ADA Negative (N=0)
Injection site reaction (General disorders) | 2 | 67 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 14 | 17 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 18 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results